CLINICAL TRIAL: NCT01956279
Title: Complementary Neurosteroid Intervention in Gulf War Illnesses (GWVI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPLD-013-12S
Record Dates: First submitted 2013-09-11; First posted 2013-10-08 (Estimated); Results first posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Fatigue; Musculoskeletal Pain; Cognitive Decline
Keywords: Pregnenolone; Gulf War Veteran; Fatigue; Musculoskeletal Pain; Cognitive Decline; Placebo Control
MeSH Terms: conditions — Fatigue; Musculoskeletal Pain; Cognitive Dysfunction | interventions — Pregnenolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pregnenolone (Arm 1) (Experimental): Pregnenolone
  Interventions: Drug: Pregnenolone
- Placebo (Arm 2) (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregnenolone — Pregnenolone 50mg BID x 14 days, followed by Pregnenolone 150 x 14 days, followed by Pregnenolone 250 mg BID x 28 days
  Arms: Pregnenolone (Arm 1)
Drug: Placebo — Placebo 50mg BID x 14 days, followed by Placebo 150 x 14 days, followed by Placebo 250 mg BID x 28 days
  Arms: Placebo (Arm 2)

SUMMARY:
This study will investigate the use of adjunctive pregnenolone for the following:

1. fatigue that has limited usual activity,
2. musculoskeletal pain involving 2 or more regions of the body and,
3. cognitive symptoms (memory, concentration, or attentional difficulties by self-report) in Veterans deployed to the Gulf War theatre of operations between 1990 and 1991.

ELIGIBILITY:
Inclusion Criteria:

* Veterans deployed to the Gulf War theatre of operations between 1990 and 1991.
* Veterans who report at least 2 of the following 3 symptoms that began in 1990 or thereafter, that lasted for more than 6 months, and that are present at the time of screening: 1) fatigue that limited usual activity, 2) musculoskeletal pain involving 2 or more regions of the body, 3) cognitive symptoms (memory, concentration, or attentional difficulties by self-report)
* Stable on medication regimen (no change in last 4 weeks) and no anticipated change in medication during study.
* Able to provide informed consent for study participation.

Exclusion Criteria:

* Subjects with a history of clinically significant neurological, metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, and/or urological disorders (e.g. unstable angina, seizures, cerebrovascular accident, decompensated congestive heart failure, central nervous system (CNS) infection, cancer [other than non-melanoma skin cancer], or history of HIV seropositivity), which would pose a risk to the patient if s/he were to participate in the study or that might confound the results of the study.
* Concurrent enrollment in another clinical trial.
* Pregnant women or women of child-bearing potential who are not surgically-sterile or not using appropriate methods of birth control.
* Use of oral contraceptives or other hormonal supplementation such as estrogen [although early studies suggested no effects on menstrual cycle, alterations in downstream metabolites or pregnenolone (such as estradiol) could theoretically impact the efficacy or oral contraceptives and/or estrogen replacement]. Similarly, it is theoretically possible that pregnenolone could be metabolized to other steroids such a DHEA, potentially resulting in hair, skin, or other steroid-related changes. Since the investigators' have determined in their prior study that pregnenolone administration does not result in downstream elevations in DHEA, DHEAS, estradiol, or testosterone, these possibilities may be unlikely.
* Women who are breast-feeding.
* Use of narcotic interventions.
* Known allergy to study medication.
* History of moderate or severe TBI (with loss of consciousness greater than 30 minutes)
* A clearly defined disease entity that accounts for the Veteran's symptoms.
* Current DSM-IV/DSM-IVTR/DSM-V diagnosis of bipolar I disorder, schizophrenia or other psychotic disorder, or dementia.
* Subjects with a DSM-IV/DSM-IVTR/DSM-V diagnosis of alcohol or substance dependence (other than nicotine or caffeine) within the last month.
* Subjects with a current suicidal or homicidal ideation necessitating clinical intervention or representing an imminent concern.
* If in the judgment of the PI it is not in the subject's best interest to participate.
* Final eligibility decisions will be determined by the PI.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine E. Marx, MD MA, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 170 participants enrolled; 142 participants were randomized after a 2-week placebo lead-in phase. The remaining 28 randomized participants were withdrawn prior to week 4 post-randomization for various reasons - including medication changes during the study (exclusionary) and participants unavailable for continued contact.
Period: Overall Study
Arm/Group | Pregnenolone (Arm 1) | Placebo (Arm 2)
Started | 82 | 88
Completed | 68 | 74
Not Completed | 14 | 14

BASELINE CHARACTERISTICS:
Population: 28 of the 170 participants were withdrawn from the study prior to reaching week 4 post-randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregnenolone (Arm 1) | Placebo (Arm 2) | Total
Number analyzed (Participants) | 82 | 88 | 170
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 81 | 88 | 169
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (5.6) | 51.4 (4.8) | 52.0 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 72 | 78 | 150
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 7
  Not Hispanic or Latino | 76 | 87 | 163
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 40 | 56 | 96
  White | 42 | 30 | 72
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 82 | 88 | 170

OUTCOME MEASURES:

1. Primary Outcome: Physical Component of the SF-36
Description: These data report changes in the mean scores in physical health symptoms at Week 8 Post-Randomization and Week 4 Post-Randomization, relative to Baseline. The SF-36 is a health survey with an 8-scale profile embedded in 36 questions that measures physical and mental components of health. Each item is scored on a 0 to 100 range, with the lowest and highest possible scores set at 0 and 100, respectively. All of these items are scored such that a high score defines a more favorable health state, and the Physical Component Score is an average of 4 of the 8 domains of the SF-36. Thus, positive changes in scores represent an improvement relative to baseline.
Time Frame: Baseline to week 4, and Baseline to week 8
Population: Change in the Physical Component Score of the SF-36. Some subjects did not reach week 8 of the study, and not all subjects completed all information at all visits.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pregnenolone (Arm 1) | Placebo (Arm 2)
Number analyzed (Participants) | 66 | 74
score on a scale
  Baseline to week 4 | 2.04 (1.50) | 2.55 (1.55)
  Baseline to week 8: number analyzed (Participants) | 55 | 60
  Baseline to week 8 | 1.23 (1.68) | 4.45 (1.75)

2. Secondary Outcome: Brief Pain Inventory (BPI)
Description: These data report changes in the mean scores in pain symptoms at Week 8 Post-Randomization and Week 4 Post-Randomization, relative to Baseline. The Brief Pain Inventory is a 14-item self-report measure designed to assess the severity, frequency and daily pattern of pain, as well as its perceived interference with quality of life. Severity is measured on a 0-10 scale with 10 being the greatest pain. Interference score is measured by a mean score of 7 items (0-10 scale) with 10 being the greatest interference. Thus, negative changes in scores represent an improvement relative to baseline.
Time Frame: Baseline to week 4, and Baseline to week 8
Population: Change in the average pain rating over the last 24 hours, and the magnitude of interference resulting from that pain. Some subjects did not reach week 8 of the study, and not all subjects completed all information at all visits.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pregnenolone (Arm 1) | Placebo (Arm 2)
Number analyzed (Participants) | 68 | 74
score on a scale
  Pain rating, Baseline to week 4: number analyzed (Participants) | 64 | 73
  Pain rating, Baseline to week 4 | -0.44 (0.14) | -0.30 (0.15)
  Pain rating, Baseline to week 8: number analyzed (Participants) | 55 | 62
  Pain rating, Baseline to week 8 | -0.09 (0.21) | -0.11 (0.22)
  Interference, Baseline to week 4: number analyzed (Participants) | 60 | 72
  Interference, Baseline to week 4 | -0.03 (0.22) | 0.00 (0.21)
  Interference, Baseline to week 8: number analyzed (Participants) | 54 | 61
  Interference, Baseline to week 8 | -0.19 (0.25) | -0.26 (0.29)

3. Secondary Outcome: Tower of London Test of the Brief Assessment of Cognition in Affective Disorders (BAC-A)
Description: These data report changes in the mean scores in cognitive symptoms at Week 8 Post-Randomization and Week 4 Post-Randomization, relative to Baseline. The Tower of London test assesses executive functioning on a scale of 0-20. (Note, if a perfect score of 20 occurs then there is the opportunity of 2 additional points, increasing the score to 22.) The higher the number, the higher the degree of executive functioning. Thus, positive changes in scores represent an improvement relative to baseline.
Time Frame: Baseline to week 4, and Baseline to week 8
Population: Change in the Tower of London Score of the BAC-A. Some subjects did not reach week 8 of the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pregnenolone (Arm 1) | Placebo (Arm 2)
Number analyzed (Participants) | 68 | 74
score on a scale
  Baseline to week 4 | 1.15 (0.37) | 1.31 (0.39)
  Baseline to week 8: number analyzed (Participants) | 56 | 63
  Baseline to week 8 | 0.98 (0.37) | 1.71 (0.41)

4. Secondary Outcome: Multidimensional Fatigue Inventory (MFI)
Description: These data report changes in the mean scores in fatigue symptoms at Week 8 Post-Randomization and Week 4 Post-Randomization, relative to Baseline. The MFI is a 20-item self-report measure designed to assess the principal manifestations of fatigue. Items are rated on a 1-5 scale indicating how true each statement was for the respondent during the last week, with some questions scored in an inverse fashion in the final calculation of the score. The 20 items are then summed, with higher scores representing greater fatigue. Thus, negative changes in scores represent an improvement relative to baseline.
Time Frame: Baseline to week 4, and Baseline to week 8
Population: Total score of the MFI-20. Some subjects did not reach week 8 of the study, and not all subjects completed all information at all visits.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pregnenolone (Arm 1) | Placebo (Arm 2)
Number analyzed (Participants) | 68 | 74
score on a scale
  Baseline to week 4: number analyzed (Participants) | 68 | 73
  Baseline to week 4 | -0.76 (1.24) | -0.27 (1.04)
  Baseline to week 8: number analyzed (Participants) | 56 | 62
  Baseline to week 8 | -3.63 (1.45) | -3.22 (1.18)

5. Secondary Outcome: Global Severity Index of the Symptom Checklist-90-Revised (SCL-90R)
Description: These data report changes in the mean scores in psychiatric symptoms at Week 8 Post-Randomization and Week 4 Post-Randomization, relative to Baseline. The SCL-90R is used as a screening measure of general psychiatric symptomatology. It includes dimensions measuring somatization, obsessive-compulsive, depression, anxiety, phobic anxiety, hostility, interpersonal sensitivity, paranoid ideation, and psychoticism. Global Severity Index (GSI) of the SCL-90R is designed to measure overall psychological distress. Higher scores reflect greater distress. This is a 90 item measure with each rated on a scale of 0-4, with 4 being the highest level of psychological distress for each item. Thus, negative changes in scores represent an improvement relative to baseline.
Time Frame: Baseline to week 4, and Baseline to week 8
Population: Average Global Severity Index score of the SCL-90. Some subjects did not reach week 8 of the study, and not all subjects completed all information at all visits.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pregnenolone (Arm 1) | Placebo (Arm 2)
Number analyzed (Participants) | 68 | 74
score on a scale
  Baseline to week 4 | -0.12 (0.04) | -0.09 (0.04)
  Baseline to week 8: number analyzed (Participants) | 56 | 63
  Baseline to week 8 | -0.16 (0.05) | -0.15 (0.05)

ADVERSE EVENTS:
Time Frame: Participants were followed for 10 weeks (or somewhat less if the participant was lost to follow-up or withdrawn during the study), with all subjects completed in a 4.5 year span.
Description: Adverse events were assessed with a structured rating scale (Hillside) every two weeks at each study visit. In addition, this structured adverse event rating scale was administered during telephone check-in assessments in between each study visit (i.e. administered weekly, either in person or by phone).
Arm/Group | Pregnenolone (Arm 1) | Placebo (Arm 2)
All-Cause Mortality (participants affected / at risk) | 1/82 | 0/88
Serious Adverse Events (participants affected / at risk) | 1/82 | 0/88
Other Adverse Events (participants affected / at risk) | 69/82 | 73/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregnenolone (Arm 1) (N=82) | Placebo (Arm 2) (N=88)
Participant death by homicide (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregnenolone (Arm 1) (N=82) | Placebo (Arm 2) (N=88)
Cold Extremities (Blood and lymphatic system disorders) | 4 | 12
Palpitations (Cardiac disorders) | 5 | 8
Tachycardia (Cardiac disorders) | 3 | 1
Tinnitus (Ear and labyrinth disorders) | 11 | 15
Blurred Vision (Eye disorders) | 10 | 19
Diarrhea (Gastrointestinal disorders) | 24 | 26
Constipation (Gastrointestinal disorders) | 12 | 17
Nausea (Gastrointestinal disorders) | 15 | 20
Vomiting (Gastrointestinal disorders) | 5 | 6
Restlessness (General disorders) | 12 | 14
Nasal Congestion (General disorders) | 20 | 33
Peripheral Edema (General disorders) | 7 | 8
Malaise (General disorders) | 6 | 2
Cramps (Musculoskeletal and connective tissue disorders) | 18 | 21
Joint Pain/Stiffness (Musculoskeletal and connective tissue disorders) | 9 | 6
Muscle Pain/Stiffness (Musculoskeletal and connective tissue disorders) | 9 | 11
Akathisia (Musculoskeletal and connective tissue disorders) | 2 | 5
Increased Motor Activity (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle Rigidity (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 1 | 1
Leg Shaking (Musculoskeletal and connective tissue disorders) | 1 | 0
Drowsiness (Nervous system disorders) | 16 | 21
Hypersomnia (Nervous system disorders) | 1 | 1
Insomnia (Nervous system disorders) | 16 | 14
Decreased Appetite (Nervous system disorders) | 9 | 14
Increased Appetite (Nervous system disorders) | 8 | 12
Dry Mouth (Nervous system disorders) | 15 | 22
Headache (Nervous system disorders) | 28 | 25
Migraine Headache (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 3 | 2
Increased Salivation (Nervous system disorders) | 5 | 5
Dizziness (Nervous system disorders) | 17 | 17
Sweating (Nervous system disorders) | 13 | 13
Decreased Interest in Sex (Nervous system disorders) | 3 | 7
Impaired Sexual Performance (Nervous system disorders) | 2 | 9
Vertigo (Nervous system disorders) | 5 | 4
Excitement / Agitation (Nervous system disorders) | 6 | 4
Confusion (Nervous system disorders) | 2 | 3
Paresthesia (Nervous system disorders) | 15 | 10
Nocturnal/Enuresis (Renal and urinary disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 3 | 2
Menstrual Disturbance (Reproductive system and breast disorders) | 3 | 4
Dermatological (Skin and subcutaneous tissue disorders) | 17 | 19
Change in Stool Color (Gastrointestinal disorders) | 0 | 1
Decreased Motor Activity (Musculoskeletal and connective tissue disorders) | 3 | 2
Pain / Stiffness (Musculoskeletal and connective tissue disorders) | 2 | 7
Disorientation (Nervous system disorders) | 4 | 3
Flatulence (Gastrointestinal disorders) | 1 | 0
Forgetfulness (Nervous system disorders) | 0 | 1
Hypertension (Cardiac disorders) | 2 | 0
Occurrence of Blank Stare (General disorders) | 1 | 0
Myoclonus (Musculoskeletal and connective tissue disorders) | 7 | 1
Rigidity (Musculoskeletal and connective tissue disorders) | 2 | 4
Fever (General disorders) | 4 | 5
Irritability (General disorders) | 8 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT01956279/Prot_SAP_000.pdf